CLINICAL TRIAL: NCT06548802
Title: Efficacy and Safety of Baricitinib in the Post-intracerebral Hemorrhage Pulmonary Injury
Acronym: BRIGHT
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University General Hospital (Other)
Collaborators: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Principal Investigator, Qiang Liu, Professor of Department of Neurology, Tianjin Medical University General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB2024-YX-067-01
Record Dates: First submitted 2024-08-07; First posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Pulmonary Injury After Intracerebral Hemorrhage
MeSH Terms: interventions — baricitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard treatment plus Baricitinib (Experimental): On standard treatment, Baricitinib was given 4mg once daily, with the first dose taken within 24 hours of the appearance of lung injury and continued for 14 days.
  Interventions: Drug: Baricitinib
- Standard treatment (No Intervention): Given standard treatment.

INTERVENTIONS:
Drug: Baricitinib — Baricitinib was given 4mg once daily, with the first dose taken within 24 hours of the appearance of lung injury and continued for 14 days.
  Arms: Standard treatment plus Baricitinib

SUMMARY:
Some patients with intracerebral hemorrhage will develop severe lung injury such as respiratory distress syndrome. Baricitinib has been approved by the FDA for severe pneumonia caused by the coronavirus, and has been used in the treatment of hospitalized patients with COVID-19. Baricitinib significantly reduced the risk of death and shortened the length of stay in COVID-19 patients. According to clinical observations, there was no significant increase in deaths or infections due to non-COVID-19 causes during recovery, nor was there a significant increase in thrombosis. Excessive inflammatory factors release can cause inflammatory storms that damage lung cells, lead to lung injury, and eventually lead to respiratory failure, respiratory distress syndrome and other conditions, endangering life safety. Studies have shown that Baricitinib can inhibit the production of excessive pro-inflammatory cytokines by lung macrophages through the JAK pathway and reduce lung injury caused by inflammatory storms. Therefore, in patients with acute stroke with lung infection or severe lung injury, short-term use of baricitinib will help to reduce lung injury and promote the recovery of neurological function, and shorten the length of hospital stay. However, there is currently a lack of effective clinical evidence of baricitinib in the treatment of lung injury after intracerebral hemorrhage, and further research is needed.

DETAILED DESCRIPTION:
The objective of this study was to evaluate the efficacy and safety of baricitinib in patients with pulmonary injury after intracerebral hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥ 18 years old;
2. The diagnosis was non-traumatic intracerebral hemorrhage, subarachnoid hemorrhage (including supratentorial deep hemorrhage, lobal hemorrhage, cerebellar hemorrhage, brainstem hemorrhage, intracerebral hemorrhage, intracerebral parenchymal hemorrhage into ventricle, subarachnoid hemorrhage), which was confirmed by CT scan.
3. Onset of ARDS within 48 hours to 7 days after admission (as defined by Berlin) : ① Patients with moderate to severe ARDS symptoms or progressive dyspnea within 7 days (100mmHg < PaO2/FiO2≤200, PEEP≥5cmH2O); ② Hypoxemia: SpO2/FiO2≤315mmHg and SpO2≤97%, and could not be explained by acute heart failure and fluid overload; ③ Need intubation or mechanical ventilation; ④ Imaging findings (chest X-ray/chest CT) : infiltration of both lungs, cannot be completely explained by pleural effusion, lobar/whole lung atelectasis and nodule;
4. There was no uncured pneumonia, interstitial lung disease, or chronic respiratory failure before the onset of the disease.
5. Able and willing to sign written informed consent and comply with the requirements of the research protocol.

Exclusion Criteria:

1. Patients diagnosed with severe intracerebral hemorrhage requiring surgical intervention with decompressive craniotomy or critically ill, near death;
2. Diagnosis of aneurysm, brain tumor, arteriovenous malformation requires surgery;
3. Recently received live or attenuated vaccine; other JAK inhibitors or other organisms are being used, or enrolled in other clinical trials;
4. Combine the following cases that are not eligible to participate in this study: ① Severe hepatic insufficiency (ALT/AST > 5xULN); ② Moderate to severe renal insufficiency (eGFR < 60ml/min/1.73m2); ③ Undergoing hemodialysis or hemofiltration; ④ Neutrophils or lymphocytes decreased (Absolute neutrophil count < 1000/ul, absolute lymphocyte count < 200/ul); ⑤ During pregnancy or childbirth;
5. Venous thromboembolism or risk of thrombosis;
6. Life expectancy after enrollment ≤24h.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-02-29 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Recovery time | From day 1 to day 30 after the lung injury occurrence.
  1. If the patient only required oxygen inhalation with the mask, SpO2≥97% of days without the mask were observed.
  2. If the patient has a tracheal intubation and ventilator-assisted breathing, observe the days needed for the patient to be removed from the ventilator.

SECONDARY OUTCOMES:
Hematoma volume after intracerebral hemorrhage | At 1, 14, and 90 days after diagnosis.
  1. CT images of the head were obtained at 1, 14, and 90 days after diagnosis. CT scan within 24 hours after diagnosis was used as the baseline analysis.
  2. If the patient is discharged from the hospital, a CT scan of the head should be performed on the 90th day if conditions permit.
NIHSS score | At 1, 3, 7, 14, 30 and 90 days after diagnosis.
  Assessed according to the National Institutes of Health Stroke Scale (NIHSS), the score ranges from 0 (asymptomatic) to 42 (death).
mRS score | At 90 days after diagnosis.
  Assessed by mRS Score on a scale of 0 (asymptomatic) to 6 (dead).
Severity score | At 1, 3, 7, 14, 30 days after diagnosis.
  Assessed by score on a scale of 0 (asymptomatic) to 8 (dead). Scores were depended on the treatment needed (Nasal tube = 1, mask = 1, non-invasive positive pressure ventilation = 1, trachea cannula = 1, glucocorticoids treatment =1, prone position ventilation = 1, ECMO= 1, death = 1.)
Murray's lung injury score | At 1, 3, 7, 14 days after diagnosis.
  The assessment was based on Murray's lung injury score.
Days without ventilator support | From diagnosis to 30 days.
  1. For patients with tracheal intubation and ventilator-assisted breathing, the tracheal intubation was removed after treatment, and only required mask oxygen inhalation or high flow oxygen inhalation days until discharge.
  2. If the patient has been discharged from the hospital and is still on no-oxygen, mask oxygen, or high-flow oxygen at the 30th day of follow-up, 30 days is recorded.
Length of ICU stay | From diagnosis to 30 days.
  1. Duration of ICU.
  2. If the patient has not reached 30 days by the time of discharge, the 30-day telephone follow-up:
     * If the patient did not continue ICU treatment, the actual number of days was recorded;
     * If the patient remains hospitalized in the ICU, 30 days is recorded.
  3. In case of death, 30 days are recorded.
APACHEⅡ score | At 1, 14, 30 days after diagnosis.
  Assessed according to acute physiology and chronic health evaluation Ⅱ (APACHEⅡ) on a scale of 0-60.
Total hospitalization days | From diagnosis to 90 days.
  Total hospitalization days.
Mortality | At 14, 30 and 90 days after diagnosis.
  Mortality of patients died because of the lung injury after ICH.
Incidence of treatment-emergent adverse events [safety and tolerability | From diagnosis to 90 days.
  Adverse events related to baricitinib are recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality, China